CLINICAL TRIAL: NCT06917170
Title: The Role of Music Therapy in Improving College Students' Mental Health and Self-efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hubei University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202211001
Record Dates: First submitted 2025-03-25; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Depressive Symptoms; Anxiety Symptoms; Stress Symptoms
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Description: Participants in this group do not receive any music therapy intervention during the study period. They continue their regular academic and daily routines.
  Intervention Type: No intervention.
- Music Therapy Intervention Group (Experimental): Description: Participants in this group receive a daily 1-hour music therapy session for 2 weeks. The intervention involves listening to rhythmically smooth, soothing music in a controlled, quiet environment. Music selection is based on evidence supporting its efficacy in reducing stress and enhancing relaxation.
  Intervention Type: Behavioral (Music Therapy).
  Interventions: Behavioral: Structured Music Therapy Program

INTERVENTIONS:
Behavioral: Structured Music Therapy Program — Description:
  Content: Participants engage in passive music therapy sessions where they listen to pre-selected music with smooth rhythms and harmonies (e.g., classical, ambient, or instrumental tracks). The music is chosen to align with evidence-based criteria for promoting relaxation and emotional regulation.
  Frequency: Daily (1 session/day).
  Duration: 1 hour per session, for a total of 14 sessions over 2 weeks.
  Setting: Conducted in a quiet, controlled environment to minimize external distractions.
  Goal: To reduce symptoms of psychological distress (depression, anxiety, stress) and enhance self-efficacy through auditory stimulation and emotional engagement.
  Arms: Music Therapy Intervention Group

SUMMARY:
Interventional Trial (Randomized Experimental Design)

Study Goal:

This clinical trial aims to evaluate the effectiveness of a structured music therapy program in improving mental health (depression, anxiety, stress) and self-efficacy among college students.

Key Questions the Study Aims to Answer:

Does music therapy significantly reduce symptoms of depression, anxiety, and stress in college students?

Does music therapy significantly enhance self-efficacy in college students?

How do improvements in mental health relate to changes in self-efficacy?

Study Design:

Researchers will compare outcomes between two groups:

Experimental Group: Receives a 2-week daily music therapy intervention (1 hour per session) in a controlled environment.

Control Group: Does not receive any music therapy intervention during the study period.

Participant Activities:

Complete pre- and post-intervention assessments using validated scales:

Depression-Anxiety-Stress Scale (DASS-21) to measure mental health status.

Self-Efficacy Scale to evaluate confidence in personal capabilities.

Experimental group participants will:

Engage in daily music therapy sessions featuring rhythmically smooth and soothing music selected to promote relaxation.

Experience the intervention in a quiet, controlled environment.

Control group participants will:

Continue their regular routines without any therapeutic intervention.

All participants will submit responses via electronic questionnaires (Wenjuanxing platform) to ensure efficient and accurate data collection.

Duration:

Intervention Period: 2 weeks.

Data Collection: Pre-intervention baseline assessment, immediate post-intervention assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be current undergraduate students (from freshmen to seniors), primarily aged between 18 and 25 years old (based on the actual age distribution of the sample).
2. Written informed consent was obtained from all participants prior to their involvement in the study.
3. Participants' baseline mental health status was not excluded (the study did not set strict clinical diagnostic criteria), but they must be able to cooperate with the intervention and complete questionnaires.

Exclusion Criteria:

1.Participants who are unable to fully participate in the 2-week intervention (such as dropping out midway or taking leave) or who do not complete the pre- and post-intervention questionnaires will be excluded.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Change in Depression, Anxiety, and Stress Scores | 2 weeks
  The assessment was conducted using the simplified version of the Depression Anxiety and Stress Scale. The full scale consists of 21 items, with each of the three subscales (depression, anxiety and stress) containing 7 items. All items are scored on a 4-point scale ranging from "0" (not applicable) to "3" (always applicable). The scores of each subscale are multiplied by 2 to obtain the score of that subscale. The higher the score, the more likely it is to indicate the presence of such emotions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei University of Science and Technology, Xianning, Hubei, China

IPD SHARING:
Plan to Share IPD: No